CLINICAL TRIAL: NCT03653208
Title: Dose Blocked-randomized, Double-blind, Placebo Controlled, Single Dose, Dose-escalation Study to Investigate the Safety, Tolerability, Pharmacokinetic Characteristics of hzVSF-v13 After Intravenous Administration in Healthy Male Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetic Characteristics of hzVSF-v13 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM_hzVSF_v13-0001
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-12

CONDITIONS: Healthy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group 1 (hzVSF-v13 10mg) (Experimental): Group 1 received a single 10mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 2 (hzVSF-v13 20mg) (Experimental): Group 2 received a single 20mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 3 (hzVSF-v13 50mg) (Experimental): Group 3 received a single 50mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 4 (hzVSF-v13 100mg) (Experimental): Group 4 received a single 100mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 5 (hzVSF-v13 200mg) (Experimental): Group 5 received a single 200mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 6 (hzVSF-v13 400mg) (Experimental): Group 6 received a single 400mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 7 (hzVSF-v13 800mg) (Experimental): Group 7 received a single 800mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Group 8 (hzVSF-v13 1200mg) (Experimental): Group 8 received a single 1200mg dose of hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13
- Placebo (Placebo Comparator): Placebo group received a single placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hzVSF-v13 — Dosage form: 10mg / 20mg / 50mg / 100mg / 200mg / 400mg / 800mg / 1200mg of hzVSF-v13 (40 mg/mL in a 5 mL vial) Frequency: Dose at Day 1 (single administration)
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: Group 1 (hzVSF-v13 10mg); Group 2 (hzVSF-v13 20mg); Group 3 (hzVSF-v13 50mg); Group 4 (hzVSF-v13 100mg); Group 5 (hzVSF-v13 200mg); Group 6 (hzVSF-v13 400mg); Group 7 (hzVSF-v13 800mg); Group 8 (hzVSF-v13 1200mg)
Drug: Placebo — Dosage form: 0.9% NaCl Solution Frequency: Dose at Day 1 (single administration)
  Other Names: 0.9% Normal saline
  Arms: Placebo

SUMMARY:
To investigate the safety/tolerability and pharmacokinetic characteristics after single intravenous (IV) administration of hzVSF-v13 (humanized Virus Suppressing Factor-variant 13) in healthy male volunteers

DETAILED DESCRIPTION:
Dose blocked-randomized, double-blind, placebo controlled, single dose, dose-escalation study to investigate the safety/tolerability and pharmacokinetic characteristics of hzVSF-v13 after IV administration in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 19 to 45 years at the time of the screening visit
* Individuals with a BMI of at least 18 kg/m2 and up to 27.0 kg/m2 weighed more than 55 kg and less than 90 kg at the time of the screening visit
* Individuals deemed clinically healthy based on medical history, physical examination, vital signs, electrocardiography (ECG), and appropriate clinical laboratory tests (provided that individuals outside the normal range may participate subject to investigator discretion)
* Individuals who have agreed to use a medically acceptable method of dual contraception and not to donate sperm from the first day until 30 days after the last day of investigational product administration
* Individuals who have voluntarily decided to participate in this clinical study and have given written consent to comply with the requirements of the study

Exclusion Criteria:

* Individuals with a clinically significant hepatic, renal, digestive, respiratory, musculoskeletal, endocrine, neurologic, psychological, hematologic, oncologic, cardiovascular, or other disease or history
* Individuals with a clinically significant history of sensitivity to the components of hzVSF-v13, drugs containing components of the same series, or other drugs (aspirin, non-steroidal anti-inflammatory drugs, antibiotics, etc.)
* Individuals testing positive in the immunogenicity test for hzVSF-v13 conducted during screening
* Individuals who have a history of drug abuse, or who turns out "positive" in test for abuse-likely drugs in the urine drug screening test
* Individuals with abnormal results for any of the following vital signs at the time of the screening visit A. Systolic blood pressure: < 90 mmHg or > 140 mmHg B. Diastolic blood pressure: < 50 mmHg or > 90 mmHg C. Heart rate: < 50 bpm or > 90 bpm
* Individuals with abnormal results for any of the following ECG items at the time of the screening visit A. PR (Pulse rate): > 210 msec B. QRS complex : > 120 msec * QRS complex is the name for the combination of three of the graphical deflections seen on a typical electrocardiogram (EKG or ECG) C. QTc (Corrected QT interval): > 450 msec
* Individuals who have participated in another clinical study or bioequivalence study in the 3 months prior to the first day of administration
* Individuals who have donated whole blood within the 2 months prior to the first day of administration, or donated blood components or received blood within the 1 month prior to the first day of administration
* Individuals who have taken barbitals or other drug-metabolizing enzyme inducers or inhibitors within the 1 month prior to screening
* Individuals who have consumed grapefruit or caffeine-containing foods within 3 days of the first administration, and individuals who are unable to avoid consuming grapefruit-containing foods from 3 days prior to admission until the date of discharge
* Individuals who have taken prescription drugs or oriental medications within 2 weeks prior to the first day of administration, or who have taken over-the-counter (OTC) drugs within the 1 week prior to the first day of administration (provided that individuals who meet other requirements may participate in the clinical study subject to investigator discretion)
* Individuals who consume high amounts of caffeine or alcohol and individuals who are heavy smokers (caffeine > 5 units/day, alcohol > 21 units/week (1 unit = 10 mL of pure alcohol), smoking > 10 cigarettes/day)
* Individuals who are unable to eat meals provided by the institution
* Individuals who have participated in the present study
* Individuals who test positive (for hepatitis B, human immunodeficiency virus (HIV), hepatitis C) on serological testing
* Individuals with veins that are not suitable for intravenous catheter insertion or multiple venipunctures
* Individuals who do not agree to use a medically acceptable method of dual contraception from the first day until 30 days after the last day of investigational product administration
* Other individuals deemed unsuitable as a subject by an investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, M.D, Principal Investigator — Seoul National University College of Medicine/Seoul National University Hospital Department of Clinical Pharmacology and Therapeutics
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (hzVSF-v13 10mg) | Group 2 (hzVSF-v13 20mg) | Group 3 (hzVSF-v13 50mg) | Group 4 (hzVSF-v13 100mg) | Group 5 (hzVSF-v13 200mg) | Group 6 (hzVSF-v13 400mg) | Group 7 (hzVSF-v13 800mg) | Group 8 (hzVSF-v13 1200mg) | Placebo
Started | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Completed | 3 | 3 | 6 | 6 | 5 | 6 | 6 | 5 | 13
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (hzVSF-v13 10mg) | Group 2 (hzVSF-v13 20mg) | Group 3 (hzVSF-v13 50mg) | Group 4 (hzVSF-v13 100mg) | Group 5 (hzVSF-v13 200mg) | Group 6 (hzVSF-v13 400mg) | Group 7 (hzVSF-v13 800mg) | Group 8 (hzVSF-v13 1200mg) | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (6.7) | 32.0 (6.6) | 32.8 (5.6) | 31.8 (4.5) | 30.3 (7.2) | 27.8 (4.9) | 35.5 (5.5) | 32.3 (5.9) | 33.4 (6.5) | 32.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Assessments by Vital Signs
Description: Systolic Blood Pressure: ≤ 90 mmHg and decrease from baseline ≥ 20 mmHg, ≥ 140 mmHg and increase from baseline ≥ 20 mmHg Diastolic Blood Pressure: ≤ 50 mmHg and decrease from baseline ≥ 10 mmHg, ≥ 90 mmHg and increase from baseline ≥ 10 mmHg Heart Rate: ≤ 40 beats/min and decrease from baseline ≥ 20 beats/min, ≥ 100 beats/min and increase from baseline ≥ 20 beats/min
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 60, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1176, 1512, 1848, 2184 hours (post-dose)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo group received placebo on Day 1 (single administration).
Arm/Group | Group 1 (hzVSF-v13 10mg) | Group 2 (hzVSF-v13 20mg) | Group 3 (hzVSF-v13 50mg) | Group 4 (hzVSF-v13 100mg) | Group 5 (hzVSF-v13 200mg) | Group 6 (hzVSF-v13 400mg) | Group 7 (hzVSF-v13 800mg) | Group 8 (hzVSF-v13 1200mg) | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13
Participants | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13

2. Secondary Outcome: Pharmacokinetic Characteristics - Cmax (Concentration Maximum)
Description: Maximum observed Concentration of hzVSF-v13 from Day1 to Day92.
Time Frame: as for outcome 1
Population: Placebo group were not included in pharmacokinetic analysis set as the it was below the quantification limit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 (hzVSF-v13 10mg) | Group 2 (hzVSF-v13 20mg) | Group 3 (hzVSF-v13 50mg) | Group 4 (hzVSF-v13 100mg) | Group 5 (hzVSF-v13 200mg) | Group 6 (hzVSF-v13 400mg) | Group 7 (hzVSF-v13 800mg) | Group 8 (hzVSF-v13 1200mg)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 5 | 6 | 6 | 5
mg/L | 1.77 (0.47) | 4.38 (1.31) | 14.04 (2.35) | 27.26 (5.82) | 45.39 (7.43) | 99.00 (14.07) | 174.43 (26.66) | 268.09 (28.07)
Statistical Analysis 1: Comparison: Group 1 (hzVSF-v13 10mg) vs Group 2 (hzVSF-v13 20mg) vs Group 3 (hzVSF-v13 50mg) vs Group 4 (hzVSF-v13 100mg) vs Group 5 (hzVSF-v13 200mg) vs Group 6 (hzVSF-v13 400mg) vs Group 7 (hzVSF-v13 800mg) vs Group 8 (hzVSF-v13 1200mg); Test type: Other; p = 0.1075, Kruskal-Wallis; Slope = 1.01

3. Secondary Outcome: PK - AUClast (Area Under the Curve Last)
Description: Area under the plasma concentration from Day1 to time of last measurable concentration.
Time Frame: as for outcome 1
Population: Placebo group were not included in pharmacokinetic analysis set as the it was below the quantification limit.
Measure: Mean (Standard Deviation); unit: h·mg/L
Arm/Group | Group 1 (hzVSF-v13 10mg) | Group 2 (hzVSF-v13 20mg) | Group 3 (hzVSF-v13 50mg) | Group 4 (hzVSF-v13 100mg) | Group 5 (hzVSF-v13 200mg) | Group 6 (hzVSF-v13 400mg) | Group 7 (hzVSF-v13 800mg) | Group 8 (hzVSF-v13 1200mg)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 5 | 6 | 6 | 5
h·mg/L | 176.74 (35.76) | 1264.31 (315.53) | 4554.13 (1143.05) | 8226.23 (2766.32) | 17386.38 (5362.11) | 39032.00 (7672.94) | 80395.46 (9269.87) | 102677.10 (25759.47)
Statistical Analysis 1: Comparison: Group 1 (hzVSF-v13 10mg) vs Group 2 (hzVSF-v13 20mg) vs Group 3 (hzVSF-v13 50mg) vs Group 4 (hzVSF-v13 100mg) vs Group 5 (hzVSF-v13 200mg) vs Group 6 (hzVSF-v13 400mg) vs Group 7 (hzVSF-v13 800mg) vs Group 8 (hzVSF-v13 1200mg); Test type: Other; p = 0.0548, Kruskal-Wallis; Slope = 1.20

ADVERSE EVENTS:
Time Frame: Up to 92 Days after dosing date (Day1).
Description: A total of 55 subjects were administered the investigational product, and a total of 52 cases of treatment emergent adverse events(TEAEs) were collected from 19 subjects (34.55%). There were no subjects that had reported serious adverse events. 4 cases of adverse events collected from 3 subjects were moderate, and all other adverse events were mild. There were no severe adverse events collected. The most common TEAE was oropharyngeal pain, 7 cases thereof were collected from 7 subjects (12.73%).
Arm/Group | Group 1 (hzVSF-v13 10mg) | Group 2 (hzVSF-v13 20mg) | Group 3 (hzVSF-v13 50mg) | Group 4 (hzVSF-v13 100mg) | Group 5 (hzVSF-v13 200mg) | Group 6 (hzVSF-v13 400mg) | Group 7 (hzVSF-v13 800mg) | Group 8 (hzVSF-v13 1200mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT03653208/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03653208/SAP_001.pdf